CLINICAL TRIAL: NCT00723541
Title: Tomosynthesis Mammography: Computer-Aided Analysis of Breast Lesions
Brief Title: Breast Lesion Analysis for Tomosynthesis Mammography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Heang-Ping Chan Ph.D, Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM 00003483; 5R01CA151443-05 (NIH)
Record Dates: First submitted 2008-07-24; First posted 2008-07-28 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Abnormal Findings on Radiological Examination of Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): Develop a computer-aided diagnostic system that will aid in the screening and detection of breast abnormalities/cancer
  Interventions: Procedure: Computer aided analysis of breast lesions

INTERVENTIONS:
Procedure: Computer aided analysis of breast lesions — Tomosynthesis mammography and computer aided analysis of breast lesions to aid in detection of breast cancer.

SUMMARY:
The purpose of this study is to develop a computer-aided diagnosis system to find breast lesions, including masses and microcalcifications, which hopefully will improve breast cancer detection and classification.

DETAILED DESCRIPTION:
The purpose of this study is to develop a computer-aided diagnosis system to find breast lesions, including masses and microcalcifications, and determine if the lesion is a cancer or not for digital tomosynthesis mammography (DTM).

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for core biopsy of a breast lesion

Exclusion Criteria:

* Pregnant females

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 872 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2016-07-12 (Actual)

PRIMARY OUTCOMES:
Achieve earlier breast cancer detection and characterization | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heang-Ping Chan, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Health System, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No